CLINICAL TRIAL: NCT04006340
Title: Comparison of Empirical and Genotypic Resistance Guided Tailored Therapy for Helicobacter Pylori Infection
Brief Title: Empirical vs Tailored Therapy for H. Pylori Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Jeong Cho, Clinical Associate Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1811-029-983
Record Dates: First submitted 2019-06-28; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Helicobacter Pylori 23S rRNA Clarithromycin Resistance Mutation; Helicobacter Pylori Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empirical group (Placebo Comparator): Patients receive conventional triple therapy containing esomeprazole 40 mg, amoxicillin 1 g and clarithromycin 500 mg twice a day for 10 days
  Interventions: Combination Product: triple therapy
- Genotypic resistance-guided tailored group (Active Comparator): Patients receive triple or quadruple therapy by resistance-associated mutations in 23S ribosomal RNA which are identified by polymerase chain reaction (PCR).
  Triple therapy contains esomeprazole 40 mg, amoxicillin 1 g and clarithromycin 500 mg twice a day for 10 days and quadruple therapy contains esomeprazole 40 mg and bismuth 300mg twice daily, tetracycline 500 mg four times daily, metronidazole 500mg three times daily for 10 days.
  Interventions: Combination Product: triple therapy; Combination Product: quadruple therapy; Diagnostic Test: dual-priming oligonucleotide-based multiplex (DPO)-PCR test

INTERVENTIONS:
Combination Product: triple therapy — esomeprazole 40 mg, amoxicillin 1 g, clarithromycin 500 mg twice a day for 10 days
Combination Product: quadruple therapy — esomeprazole 40 mg and bismuth 300mg twice daily, tetracycline 500 mg four times daily, metronidazole 500mg three times daily for 10 days
  Arms: Genotypic resistance-guided tailored group
Diagnostic Test: dual-priming oligonucleotide-based multiplex (DPO)-PCR test — Resistance of clarithromycin 23S rRNA point mutation
  Arms: Genotypic resistance-guided tailored group

SUMMARY:
We aimed to compare the efficacy of genotypic resistance-guided tailored therapy vs empirical therapy for eradication of Helicobacter pylori (H. pylori) infection in randomized controlled trials.

DETAILED DESCRIPTION:
Empirical therapy is conventional triple therapy (proton pump inhibitor (PPI) standard dose, amoxicillin 1 g and clarithromycin 500 mg twice a day for 10 days). Genotypic resistance-guided tailored therapy is the method which is chosen by DPO-PCR test. While the patients who have positive result of clarithromycin resistance receive the quadruple therapy(PPI standard dose, bismuth 300mg twice daily, tetracycline 500 mg four times daily, metronidazole 500mg three times daily for 10 days), clarithromycin susceptible patients receive the triple therapy.

H. pylori is difficult to cultivate, cultivation of H. pylori and minimum inhibitory concentration test as a resistance test method are very difficult and take a long time. Recently, tailored treatment based on clarithromycin susceptibility has been proposed by dual-priming oligonucleotide-based multiplex (DPO)-PCR test. This is a method to confirm the mutation of A2142G and A2143G by PCR, which are known to be highly related to the resistance of clarithromycin 23S rRNA point mutation. This test is performed only by gastric biopsy. The examination time is also short as several hours, and sensitivity and specificity are about 80-85%.

Antibiotic resistance of H. pylori, especially clarithromycin resistance, is a cause of major failure of its eradication, and Korea 's clarithromycin resistance rate is reported to be about 37%. The eradication rate of standard triple therapy reported in Korea is also unsatisfactory as antibiotic resistance rate of H. pylori increases. The ideal eradication rate for H. pylori is approximately 90%, but in the meta-analysis of the recently reported primary eradication, the overall eradication rate was 74.6% in the intention to treat analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with H. pylori who had undergone endoscopic resection for gastric neoplasm
* Patients with H. pylori who had diagnosed at peptic ulcer disease, MALT lymphoma

Exclusion Criteria:

* history of gastrectomy
* patients aged younger than 20 years or older than 80 years
* history of H. pylori eradication therapies or other antibiotics therapy within a month
* previous allergic reaction to the study drugs (amoxicillin, clarithromycin, metronidazole, tetracycline, and esomeprazole)
* contraindication to treatment drugs
* pregnant or lactating women
* severe concurrent illness

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2019-01-04 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-08-31 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | 13C-UBT at least 4 weeks after completion of treatment
  Eradication rate of H. pylori infection

CONTACTS AND LOCATIONS:
Overall Officials: Soo-Jeong Cho, M.D., ph.D., Principal Investigator — Department of Internal Medicine and Liver Research Institute,
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim JL, Cho SJ, Chung SJ, Lee A, Choi J, Chung H, Kim SG. Empiric Versus Clarithromycin Resistance-Guided Therapy for Helicobacter pylori Based on Polymerase Chain Reaction Results in Patients With Gastric Neoplasms or Gastric Mucosa-Associated Lymphoid Tissue Lymphoma: A Randomized Controlled Trial. Clin Transl Gastroenterol. 2020 Sep;11(9):e00194. doi: 10.14309/ctg.0000000000000194. PMID 33094958